CLINICAL TRIAL: NCT03775785
Title: Effect of Targeted vs Standard Fortification of Breast Milk on Growth and Development of Preterm Infants (≤ 32 Weeks): a Randomised Controlled Trial
Brief Title: Targeted vs Standard Fortification of Breast Milk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Princess Anna Mazowiecka Hospital, Warsaw, Poland (Other)
Collaborators: Medical University of Warsaw (Other); Institute of Mother and Child (Unknown)
Responsible Party: Principal Investigator, Joanna Seliga-Siwecka, Principal Investigator, Princess Anna Mazowiecka Hospital, Warsaw, Poland
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1/2018
Record Dates: First submitted 2018-12-10; First posted 2018-12-14 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-12

CONDITIONS: BPD - Bronchopulmonary Dysplasia; NEC - Necrotizing Enterocolitis; Weight Gain; VLBW - Very Low Birth Weight Infant; ROP - Retinopathy of Prematurity
Keywords: enteral nutrition; fortification; tailored enteral nutrition
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Enterocolitis, Necrotizing; Weight Gain; Retinopathy of Prematurity

STUDY DESIGN:
Intervention Model Description: This is a multi-centre superiority randomised parallel group, 1:1 allocation study.
  After reaching 80 ml/kg/day of enteral feeding, patients will be randomised to receive standard fortification-SF (Bebilon HMF, Nutricia) or targeted fortification -TF (proteins, lipids,carbohydrates). Allocation will be performed electronically.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The decision to start fortification will be made by the attending physician blinded to the intervention allocated. An employee outside the research team will feed data into the computer in separate datasheets so that the researchers can analyse data without having access to information about the allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tailored enteral nutrition (Experimental): Tailored Human milk fortification procedure Tailored milk fortification will be done twice a day (8 am and 8 pm) for each following 12 hour nursing shift. Standard fortification will be added first. The remainder amount of protein, lipids and carbohydrates required to meet the recommended by ESPGHAN doses will be acheived by adding single ingrediant nutrients.
  Interventions: Dietary Supplement: Tailored enteral nutrition
- standard enteral nutrition (No Intervention): Standard fortification will be added according to the unit protocol.

INTERVENTIONS:
Dietary Supplement: Tailored enteral nutrition — The mean of three measurements per batch (3 x 2-3ml) will be used to calculate the required amount of extra fat, protein, and carbohydrate for the following 3 days of fortification using a predefined Excel spread sheet (Microsoft Inc, Redmond, Washington).
  The intervention will consist of adding fat, protein, and/or carbohydrate to achieve target levels of macronutrients.
  The defined macronutrient concentration in breast milk is 4.4 g/100 mL of fat, 3 g/100 mL of protein, and 8.8 g/ 100 mL of carbohydrate to meet the European Society for Paediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN) guidelines (6.6 g/kg/d of fat, 4.5 g/kg/d of protein, and 13.2 g/kg/d of carbohydrate) assuming an intake of 150 mL/kg/d.
  Arms: tailored enteral nutrition

SUMMARY:
BACKGROUND:

Human milk (HM) is recommended for all very low birth infants (VLBW)). Breast-milk is highly variable in nutrient content, failing to meet the nutritional demands of VLBW. Fortification of HM is recommended to prevent extra-uterine growth retardation and associated poor neurodevelopmental outcome. However, standard fortification with fixed dose multicomponent fortifier does not account for the variability in milk composition. Targeted fortification is a promising alternative and needs further investigation.

The aim of the study is to evaluate if targeted fortification of human milk may optimize growth and development in preterm infants.

STUDY DESIGN:

Randomized single blind controlled trial.

METHODS & ANALYSIS:

We will recruit preterm infants (≤ 32 weeks of gestation) within the first 7 days of life. After reaching 80 ml/kg/day of enteral feeding, patients will be randomised to receive standard fortification (HMF, Nutricia) or targeted fortification (modular components: Bebilon Bialko, Nutricia - protein, Fantomalt, Nutricia - carbohydrates, Calogen, Nutricia - lipids). The intervention will continue until 37 weeks of post-conception age, or hospital discharge. Parents and outcome assessors will be blinded to the intervention.

The primary outcome - weight gain velocity will be measured starting from the day infants regain their birth weight up to 4 weeks, then weekly until discharge.

Secondary outcomes such as neurodevelopment at 12 months of corrected age (CA) will be assessed with Bayley Scale of Development III, repeated at 36 months of CA. Additionally a Wescheler Preschool and Primary Scale of Intelligence IV test will be applied at 3,5 years of CA. Secondary outcomes such as length and head growth, body composition will be assesed at discharge and at 4 months. Incidence of necrotizing enterocolitis (NEC), sepsis, retinopathy of prematurity (ROP) and bronchopulmonary dysplasia (BPD) will also be followed.

DETAILED DESCRIPTION:
Study design and setting This is a multi-centre superiority randomised parallel group, 1:1 allocation study. Patients will be recruited at three departments of neonatology and intensive care units: Department of Neonatology and Neonatal Intensive Care, Division of Neonatal Intensive Care (Medical University of Warsaw), and the Institute of Mother and Child. Follow up will be carried out at the Department of Paediatrics.

The study is lead by the Department of Neonatology and Neonatal Intensive Care (KAROWA) with approximately 3000 (100 ≤ 32 weeks of gestation) deliveries per year and 12 intensive care and 40 high dependency neonatal beds.

Recruitment Recruitment will take place between June 2019 and December 2020. Parents of infants born at less than 32 weeks of gestation will be approached within the first week of life.

Randomisation After reaching 80 ml/kg/day of enteral feeding, patients will be randomised to receive standard fortification (SF) or targeted fortification (TF) (proteins, lipids, carbohydrates). Allocation will be performed electronically.

Interventions Human milk fortification procedure Milk fortification will be done twice a day (8 am and 8 pm) for each following 12 hour nursing shift (Appendix 1).

A 10 mL aliquot from each batch of native breast milk will be used for macronutrient analysis using a human milk analyser Miris® as per protocol. The remaining batch will first be fortified with the standard fortifier. Macronutrient analysis will determine how much extra fat, protein, and/or carbohydrate is needed to obtain target fortified breast milk.

An experienced laboratory technician will perform milk analysis in the neonatal intensive care unit (NICU) research laboratory at KAROWA twice per week at 10:00 am (Monday/Friday) from batches collected from the two previous days. Milk samples from other sites will be delivered by medical transport in secure freezing containers at 8:00 am.

The mean of three measurements per batch (3 x 2-3ml) will be used to calculate the required amount of extra fat, protein, and carbohydrate for the following 3 days of fortification using a predefined Excel spread sheet (Microsoft Inc, Redmond, Washington). Milk analysis will be performed in both treatment arms; however only the intervention group will receive TF. Results, together with required amounts of macronutrients, will be emailed to the participating centres before noon the same day.

The defined macronutrient concentration in breast milk is 4.4 g/100 mL of fat, 3 g/100 mL of protein, and 8.8 g/ 100 mL of carbohydrate to meet the European Society for Paediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN) guidelines (6.6 g/kg/d of fat, 4.5 g/kg/d of protein, and 13.2 g/kg/d of carbohydrate) assuming an intake of 150 mL/kg/d.

Target fortification will be done in 3 steps:

1. Determination of macronutrients concentration in own mothers´s milk (OMM)/human donor milk (HDM).
2. Standard fortification (SF) (human milk fortifier - HMF).
3. Targeted fortification (TF): adding fat, protein, and/or carbohydrate to achieve target levels of macronutrients.

In cases where a macronutrient component after SF will exceed the target value, only the other deficient macronutrient components will be adjusted.

Safety Prescription of TF will be completed before noon. Bedside nurses will prepare batches of fortified breast milk including the additives for TF.

Data from breast milk analyses, fortification, and enteral intake will be documented daily. Acid base status, blood urea nitrogen (BUN), and glucose will be determined as per NICU routine.

The intervention will continue until 37 weeks of post-conception age, or hospital discharge. Parents and outcome assessors will be blinded to the intervention.

Randomization A study number together with the allocated treatment will be assigned by the platform. Patient's data along with the result of the allocation will be sent to statistical team. The randomisation list will remain with the statistical team for the whole duration of the study. Randomisation will be conducted without any influence of the principal investigators, clinicians, recruitment or follow up staff.

Blinding The decision to start fortification will be made by the attending physician blinded to the intervention allocated. An employee outside the research team will feed data into the computer in separate datasets so that the researchers can analyse data without having access to information about the allocation.

Sample size The sample size required to compare two means in two-sided equality test was estimated based on results from a prior double blind, randomised clinical trial, investigating the effect of target fortification vs standard fortification of breast milk on the changes of anthropometric parameters and body composition in preterm children. It was determined, that a mean difference of weight gain 1.9 g/kg/day between groups would be clinically important and feasible during intervention. between the study groups with a power of 80% and α=0.05, a sample of 91 infants is needed in each study group. Allowing for 10% of loss to follow-up, the target number of 200 premature infants will be recruited.

ELIGIBILITY:
Inclusion Criteria:

Patients eligible for the trial must comply with all of the following at randomization:

1. Gestational age at birth ≤ 32 weeks
2. Enteral feeding of at least 80ml/kg/day
3. Donor or maternal milk based enteral feeding (at least 50%)
4. Parenteral/legal guardian consent

Exclusion Criteria:

1. >50% formula based enteral feeding
2. Small for gestational age (birth weight < 3rd percentile)
3. Congenital abnormalities which increase the risk of NEC
4. NEC
5. Withdrawal of feeding > 7 days
6. Sepsis
7. Death

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Growth | from birth at postmentrual age <32 to up to 37 weeks of post-conceptional age
  weight will be assessed every day.
Velocity of weight gain in grams | from birth at postmentrual age <32 to up to 37 weeks of post-conceptional age
  weight will be assessed every day.

SECONDARY OUTCOMES:
Neurodevelopmental outcome | at 12 and 36 weeks of corrected age.
  the number of infants with mental development index (MDI) Bayley Scale of Development III
Necrotizing enterocolitis (NEC) | from birth at postmentrual age <32 to up to 37 weeks of post-gestational age
  The number of patients NEC >1 stage as defined by Bell's criteria
Bronchopulmonary dysplasia (BPD) | from 28 days at postmentrual age <32 to up to 37 weeks of post gestational age
  The number of patients with (BPD) defined as oxygen requirement of > 21% at 28 days of life
Late onset sepsis (LOS) | from 72 hours of life at postmentrual age <32 up to 37 weeks of post gestational age
  The number of patients with LOS defined as a positive blood culture or a positive cerebral spinal fluid culture
Retinopathy of prematurity (ROP) | from 3 weeks of life at postmentrual age <32 to 37 weeks of post gestational age
  The number of patients with ROP > grade I as defined as the World Health Organisation criteria

CONTACTS AND LOCATIONS:
Locations (2):
- Poland (2):
  - Department of Neonatology and Neonatal Intensive Care Warsaw Medical University, Warsaw
  - Division of Neonatology and Neonatal Intensive Care, 1st Department of Obstetrics and Gynaecology, The Medical University of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participation data will be available on request from the corresponding author. Data reuse will be permitted for meta-analysis.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 24 months after data analysis completion.
Access Criteria: researchers

REFERENCES:
- [Derived] Seliga-Siwecka J, Chmielewska A, Jasinska K. Effect of targeted vs standard fortification of breast milk on growth and development of preterm infants (</= 32 weeks): study protocol for a randomized controlled trial. Trials. 2020 Nov 23;21(1):946. doi: 10.1186/s13063-020-04841-x. PMID 33225961